CLINICAL TRIAL: NCT03704662
Title: A Randomized, Phase II Clinical Trial of Preoperative Fractionated Radiation Therapy Versus Stereotactic Body Radiation Therapy for Resectable or Borderline Resectable, or Locally Advanced Type A Pancreatic Adenocarcinoma
Brief Title: Preoperative Fractionated Radiation Therapy Versus Stereotactic Body Radiation Therapy for Resectable or Borderline Resectable, or Locally Advanced Type A Pancreatic Adenocarcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William Hall, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00033061
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
Keywords: resectable pancreatic adenocarcinoma; borderline resectable pancreatic adenocarcinoma; Stereotactic Body Radiation Therapy; Preoperative Fractionated Radiation Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Radiosurgery; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stereotactic Body Radiation Therapy (Other): Patients undergo Stereotactic Body Radiation Therapy (25 to 35 Gy over five fractions)
  Interventions: Radiation: Stereotactic Body Radiation Therapy
- Preoperative Fractionated Radiation Therapy and Chemotherapy (Other): Concurrent chemotherapy with radiation treatment (50.4 Gy over 28 fractions).
  Interventions: Radiation: Preoperative Fractionated Radiation Therapy and Chemotherapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SBRT
  Arms: Stereotactic Body Radiation Therapy
Radiation: Preoperative Fractionated Radiation Therapy and Chemotherapy — Conventional concurrent chemotherapy and radiation therapy.
  Arms: Preoperative Fractionated Radiation Therapy and Chemotherapy

SUMMARY:
Patients are randomized into two arms. Arm A patients will receive Stereotactic Body Radiation Therapy (SBRT) and Arm B patients with receive conventional concurrent chemotherapy and radiation therapy.

DETAILED DESCRIPTION:
RATIONALE: There are limited studies comparing novel radiation treatments with stereotactic body radiation therapy (SBRT) in pancreatic adenocarcinoma to conventional fractionation. Much of the existing literature indicates this technique is safe and convenient for patients, as compared with conventionally fractionated concurrent chemo-radiation therapy. However, there has been no direct comparison of these two treatment modalities when given in the preoperative setting. It also remains uncertain if SBRT results in similar nodal downstaging to preoperative, conventionally fractionated chemo-RT.

STUDY DESIGN: This study is a prospective, open-label, randomized, parallel, two-arm, phase II clinical trial. Patients meeting the eligibility criteria will be randomized after a minimum of one cycle of induction chemotherapy. These patients will be required to have no biopsy-proven distant disease on repeat staging studies before randomization. Patients who have radiologically equivocal evidence of distant metastatic disease (small lung nodules, or liver lesions that cannot be definitively characterized, etc.) are also eligible for enrollment. Patients with biopsy-proven metastatic disease are not eligible. The total number of patients planned for accrual is approximately 102 patients (51 patients per arm), with 14 additional patients enrolled to account for a roughly 15% drop out rate.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically confirmed (histologic or cytological), resectable, borderline resectable, or locally advanced type A adenocarcinoma of the pancreas; patients must have resectable, borderline resectable, or locally advanced type A disease, based on institutional standardized criteria and tumor board review.
2. Patients with and without regional adenopathy are eligible.
3. Patients are eligible with either no evidence of distant metastatic disease, or "equivocal" evidence of distant metastatic disease, as judged by multidisciplinary review. This "equivocal" definition can include small lung or liver lesions that are not able to be radiographically characterized otherwise. Any biopsy-proven metastatic disease will make the patient ineligible for study participation.
4. History/physical examination, including collection of weight and vital signs, within 45 days prior to start of treatment.
5. Diagnostic abdominal/pelvic CT with IV contrast or abdominopelvic MRI scan with perfusion and diffusion-weighted sequences within 45 days prior to study entry.
6. Chest CT scan or X-ray within 30 days prior to study entry.
7. Radiation treatment planning abdominal CT. A recommended abdominal MRI will be done as a simulation (SIM) with interpretation. The CT SIM will not be done with interpretation. Positron emission tomography (PET) scan and MRI are both optional but encouraged. Ability to undergo abdominal MR scans for staging and radiation planning and follow-up is optional but encouraged.
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2 within 14 days of randomization.
9. Age ≥ 18.
10. Heme Onc (Chem 24) and cancer antigen (CA) 19-9/carcinoembryonic antigen (CEA) within 45 days prior to treatment, as follows:

    * Absolute neutrophil count (ANC) ≥ 1,000 cells/mm3
    * Platelets ≥100,000 cells/mm3 (see section 4)
    * Hemoglobin ≥ 8.0 g/dl (Note: The use of transfusion or other intervention to achieve Hgb ≥ 8.0 g/dl is acceptable.)
    * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) < 4 x upper limit of normal
    * Total bilirubin < 1.5 x upper normal mg/dL
    * Alkaline phosphatase < 4 x upper limit of normal
11. Not on hemodialysis.
12. Negative serum pregnancy test (if applicable).
13. Ability to swallow oral medications.
14. Patients must have had at least one cycle of systemic chemotherapy without evidence of distant progression.
15. Patient must provide study-specific informed consent prior to study entry.
16. Women of childbearing potential and male participants who are sexually active must practice adequate contraception.

Exclusion Criteria:

1. Distant metastatic disease.
2. Prior invasive malignancy (except nonmelanomatous skin cancer), unless disease free for a minimum of three years (for example, carcinoma in situ of the breast, oral cavity or cervix are all permissible).
3. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation therapy fields.
4. Any major surgery within 28 days prior to study entry (for example, insertion of a vascular access device or biliary stent, exploratory laparotomy and/or laparoscopy are not considered major surgery; biliary or gastric bypass is considered major surgery).
5. Severe, active comorbidity, defined as follows:

   * Unstable angina and/or congestive heart failure requiring hospitalization within the last six months.
   * Transmural myocardial infarction within three months prior to study entry.
   * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration.
   * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy within 30 days before registration.
   * Uncontrolled malabsorption syndrome significantly affecting gastrointestinal function.
   * Any unresolved bowel or bile duct obstruction.
   * Major resection of the stomach or small bowel that could affect the absorption of capecitabine.
   * Acquired immune deficiency syndrome (AIDS), based upon current Center for Disease Control (CDC) definition. Note, however, that HIV testing is not required for entry into this protocol. The need to exclude patients with AIDS from this protocol is necessary because patients receiving antiretroviral therapy may experience possible pharmacokinetic interactions with capecitabine.
   * Absence of any significant medical comorbidity which would preclude the consideration of major pancreatic surgery.
6. Pregnancy or women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception during the course of the study and for women three months after study therapy is completed and for men six months after study therapy is completed. This exclusion is necessary because the treatment involved in this study may be significantly teratogenic.
7. Women who are lactating at the time of registration and who plan to be lactating through three months after study therapy is completed.
8. Prior allergic reaction to capecitabine or gemcitabine.
9. Participation in another interventional clinical treatment trial while on study (observational trials are permitted).
10. Patients taking nonprotocol-specified chemotherapy agents or immune modulating agents for other medical conditions are not permitted to participate in this trial. Any medication questions should be reviewed by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2018-10-22 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of subjects who present with node-positive disease following surgical resection. | 8 weeks postradiation
  Subjects will undergo surgical resection within three to eight weeks following treatment.

CONTACTS AND LOCATIONS:
Overall Officials: William Hall, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No